CLINICAL TRIAL: NCT01479062
Title: Multi-Channel Automated Diet and Physical Activity Intervention for Pre-Diabetics (ALIVE-PD)
Brief Title: Multi-Channel Automated Diet and Physical Activity Intervention for Pre-Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berkeley Analytics, Inc. (Industry)
Collaborators: Palo Alto Medical Foundation (Other)
Responsible Party: Principal Investigator, Gladys Block, Principal Investigator, Berkeley Analytics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R44NR012617-01 (NIH)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2016-07

CONDITIONS: Pre-diabetes; Diabetes; Obesity
Keywords: behavior change; pre-diabetes; prevention; diabetes prevention; Hemoglobin A1c; glucose; physical activity; nutrition; email; web; obesity
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- participation in Alive-PD (Experimental): Alive-PD lifestyle intervention with multi-channel delivery
  Interventions: Behavioral: Alive-PD
- Control (Placebo Comparator): Usual care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Alive-PD — Weekly email/web goal-setting intervention to improve physical activity, diet and weight loss for pre-diabetics, with additional phone support
  Arms: participation in Alive-PD
Behavioral: Usual Care — Placebo Control
  Arms: Control

SUMMARY:
The trial will test whether the Alive multi-channel delivery health behavior program can positively affect weight and glucose level in pre-diabetics.

ELIGIBILITY:
Inclusion Criteria:

* at least one measurement in past 2 yrs of fasting plasma glucose of 100-125 mg/dl or impaired glucose tolerance
* at least one measurement of body mass index (BMI) >=27 in the past two years
* age 40-79
* no use of diabetes medications within the past two years
* member of Kaiser Permanente of Northern California (KPNC) for at least 2 years
* live in a 25 mile radius of the KPNC Research Clinic in Oakland, CA

Exclusion Criteria:

* comorbidities that would contraindicate the gradual adoption of light/moderate physical activity, such as a recent cardiovascular event, severe chronic obstructive pulmonary disease, advanced arthritis, or poorly controlled hypertension

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body weight | at 3 months, 6 months and one year
  Mean weight loss and the proportion of subjects who achieve a 5% body weight loss at 3 and 6 months and maintain at 12 months
Change from baseline in diabetes risk markers | at 3 months, 6 months and one year
  Change in blood glucose level and hemoglobin A1c (HbA1c) as measured in clinic at 3 and 6 months and maintain at 12 months

SECONDARY OUTCOMES:
Change from baseline in physical activity and dietary factors | 3 months and 12 months
  Extent of change in physical activity and dietary factors as reported in questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Gladys Block, PhD, Principal Investigator — Berkeley Analytics, Inc.
Locations (1):
- Palo Alto Medical Foundation Research Institute, Palo Alto, California, United States

REFERENCES:
- [Background] Block G, Azar KM, Block TJ, Romanelli RJ, Carpenter H, Hopkins D, Palaniappan L, Block CH. A Fully Automated Diabetes Prevention Program, Alive-PD: Program Design and Randomized Controlled Trial Protocol. JMIR Res Protoc. 2015 Jan 21;4(1):e3. doi: 10.2196/resprot.4046. PMID 25608692
- [Result] Block G, Azar KM, Romanelli RJ, Block TJ, Hopkins D, Carpenter HA, Dolginsky MS, Hudes ML, Palaniappan LP, Block CH. Diabetes Prevention and Weight Loss with a Fully Automated Behavioral Intervention by Email, Web, and Mobile Phone: A Randomized Controlled Trial Among Persons with Prediabetes. J Med Internet Res. 2015 Oct 23;17(10):e240. doi: 10.2196/jmir.4897. PMID 26499966